CLINICAL TRIAL: NCT01040910
Title: A Double Blind Placebo Controlled Study of Cannabis Smoking in Inflammatory Bowel Disease
Brief Title: Cannabis for Inflammatory Bowel Disease
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, NAFTALI TIMNA, MD, Meir Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: cannabis1
Record Dates: First submitted 2009-12-29; First posted 2009-12-30 (Estimated); Last update posted 2011-12-16 (Estimated); Status verified 2011-12

CONDITIONS: Crohn's Disease; Ulcerative Colitis
Keywords: cannabis; Crohn's disease; Ulcerative colitis; IBD
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Marijuana Abuse

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- cannabis smoking for IBD (Active Comparator): patients with active disease receiving active cannabis for smoking
  Interventions: Drug: smoking of cannabis
- patients smoking non active cannabis (Placebo Comparator): patients with active disease receiving cannabis from which active ingredients have been chemically removed
  Interventions: Drug: smoking cigarettes with placebo

INTERVENTIONS:
Drug: smoking of cannabis — smoking of cannabis, 2 cigarettes a day, equivalent to about 50 mg THC
  Arms: cannabis smoking for IBD
Drug: smoking cigarettes with placebo — smoking cigarettes with cannabis that was chemically treated so that most active ingredients were removed
  Arms: patients smoking non active cannabis

SUMMARY:
Background: The marijuana plant Cannabis has been used for centuries in the medicinal treatment of many disorders and is still the subject of medical research and public debate. Cannabinoids have been purported to alleviate a variety of neurological conditions such as MS-related symptoms including spasticity, pain, tremor and bladder dysfunction. Other neurological conditions like chronic intractable pain, dystonic movement disorders and Tourette's Syndrome were all reported to be alleviated by cannabis use. Cannabis has been used to treat anorexia in AIDS and cancer patients. In gastroenterology cannabis has been used to treat symptoms and diseases including anorexia, emesis, abdominal pain, gastroenteritis, diarrhoea, intestinal inflammation and diabetic gastroparesis.

Cannabinoids have also a profound anti inflammatory effect, mainly through the CB2 receptor. Cell mediated immunity may be impaired in chronic marijuana users. And a potent anti-inflammatory effect of cannabis was observed in rats . Studying the functional roles of the endocannabinoid system in immune modulation reveals that there are no major immune events which do not involve the endocannabinoid system. Cannabinoids shift the balance of pro-inflammatory cytokines and anti-inflammatory cytokines towards the T-helper cell type 2 profiles (Th2 phenotype), and suppress cell-mediated immunity whereas humoral immunity may be enhanced. They are therefore used for various inflammatory conditions including rheumatoid arthritis and asthma. In a mouse model of colitis cannabinoids were found to ameliorate inflammation and there are many anecdotal reports about the effect of cannabis in inflammatory bowel disease. However, there are no methodical reports of the effect of cannabis on inflammatory bowel disease. The aim of the proposed study is to examine in a double blind placebo controlled fashion the effect of smoking cannabis on disease activity in patients with IBD.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a diagnosis IBD at least 3 months before recruitment will be eligible to the study.
2. Patients with active disease who are resistant to either 5 ASA, steroids or immunomodulators, or who can not receive those drugs due to adverse reactions will be offered the possibility of smoking cannabis at a dose of two cigarettes a day which will contain either regular cannabis or pre treated cannabis as placebo.
3. Disease activity index of either CDAI of more then 200 in Crohn's disease or Mayo score above 3 in UC.
4. Age above 20.

Exclusion Criteria:

1. Patients with a known mental disorder
2. Patients who are deemed to be at a high risk of abuse or addiction to the study drug.
3. Pregnant women
4. Patients who are sensitive to any of the ingredients of the study medication.
5. Patients who are unable to give informed consent.
6. Patients who may need surgery in the near future.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-01; Primary Completion 2012-06 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
reduction of CDAI by 70 points | 8 weeks

SECONDARY OUTCOMES:
adverse events due to cannabis smoking | 8 weeks
change in quality of life before and at the end of study | 8 weeks
change in IL-10. IL-2. TGF beta | week 0 and week 8

CONTACTS AND LOCATIONS:
Overall Officials: Fred Konikoff, professor, Study Chair — Sackler school of medicine Tel Aviv university; Timna Naftali, Principal Investigator — Meir Medical Center
Locations (2):
- Israel (2):
  - Meir hospital, Kfar Saba
  - Meir Medical center, Kfar Saba

REFERENCES:
- [Derived] Naftali T, Bar-Lev Schleider L, Scklerovsky Benjaminov F, Konikoff FM, Matalon ST, Ringel Y. Cannabis is associated with clinical but not endoscopic remission in ulcerative colitis: A randomized controlled trial. PLoS One. 2021 Feb 11;16(2):e0246871. doi: 10.1371/journal.pone.0246871. eCollection 2021. PMID 33571293
- [Derived] Naftali T, Bar-Lev Schleider L, Dotan I, Lansky EP, Sklerovsky Benjaminov F, Konikoff FM. Cannabis induces a clinical response in patients with Crohn's disease: a prospective placebo-controlled study. Clin Gastroenterol Hepatol. 2013 Oct;11(10):1276-1280.e1. doi: 10.1016/j.cgh.2013.04.034. Epub 2013 May 4. PMID 23648372